CLINICAL TRIAL: NCT04961320
Title: Assessing Efficacy of an Occupational Therapy Fatigue Management-Based Intervention for Patients With Metastatic Renal Cell Carcinoma
Brief Title: Occupational Therapy Fatigue Management-Based Intervention for Metastatic Renal Cell Carcinoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20566; NCI-2021-05561 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20566 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-07-14 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Renal Cell Carcinoma; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (OT, questionnaires) (Experimental): Patients participate in OT sessions weekly for 3 weeks over 30 minutes each. Patients also complete questionnaires to assess anxiety, depression, fatigue and pain at baseline, 5 and 12 weeks.
  Interventions: Behavioral: Occupational Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Occupational Therapy — Participate in OT session
  Other Names: OT
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial studies the effects of occupational therapy fatigue management in patients with renal cell cancer that has spread to other places in the body (metastatic). Many patients diagnosed with cancer experience cancer-related fatigue. These patients that are also on immunotherapy can experience added distressing fatigue that impacts their daily lives. Occupational therapy uses a client-centered and holistic approach to work collaboratively with patients to assess fatigue and develop strategies to manage each individual's specific needs. Fatigue-based management is a fundamental component of occupational therapy rehabilitation regimens. This trial may help patients address and reduce their fatigue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if an occupational therapy (OT)-based intervention can reduce cancer-related fatigue by 10 percent as measured by the brief fatigue inventory (BFI) tool, in patients undergoing immunotherapy for metastatic renal cell carcinoma.

SECONDARY OBJECTIVES:

I. To determine if an OT-based intervention can improve pain ratings. II. To determine if an OT-based intervention can improve indices of depression. III. To determine if an OT-based intervention can improve indices of anxiety. IV. To determine if an OT-based intervention can maintain a reduced level of fatigue beyond the period of intervention.

OUTLINE:

Patients participate in OT sessions weekly for 3 weeks over 30 minutes each. Patients also complete questionnaires to assess anxiety, depression, fatigue and pain at baseline, 5 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over.
* Sufficiently fluent in English.
* Cytologically or pathologically verified diagnosis of renal cell carcinoma (RCC).
* Evidence of metastatic disease.
* Clinician assessed prognosis of greater than or equal to six months.
* Patients who are undergoing immunotherapy treatment (with a checkpoint inhibitor) for advanced kidney cancer who have grade 1 or 2 fatigue based on physician assessment at the time of study entry.
* Willing and independently able to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue Inventory Score | Baseline up to 5 weeks
  Percentage of patients with a 10 percent or greater reduction in brief fatigue inventory score.
  Brief Fatigue Inventory is scored on an 10 points scale (0 to 10), with higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
Pain ratings | Baseline up to 5 and 12 weeks
  Pairwise differences of score will be calculated for the PAIN assessment tools per patient, between baseline and the follow-up time points of 5 and 12 weeks. Descriptive statistics will be used to summarize the change in pain score, (from baseline to 5- and 12- weeks). Plots will be utilized to help visualize the changes in scores over time. The scale for the PAIN tool ranges 0-10, with the higher scores indicating worse outcomes.
Depression | From baseline to 5 and 12 weeks
  Pairwise differences of score will be calculated for the Depression assessment tool per patient, between baseline and the follow-up time points of 5 and 12 weeks. Descriptive statistics will be used to summarize the change in the PROMIS Depression score, (from baseline to 5- and 12- weeks). Plots will be utilized to help visualize the changes in Depression scores over time. Total score for the PROMIS Depression tool ranges from 8 to 40, with higher scores indicating worse outcomes.
Anxiety | From baseline to 5 and 12 weeks
  Pairwise differences of score will be calculated for the PROMIS Anxiety tool per patient, between baseline and the follow-up time points of 5 and 12 weeks. Descriptive statistics will be used to summarize the change in the anxiety score, indices of anxiety and depression, and fatigue score (from baseline to 5- and 12- weeks). Plots will be utilized to help visualize the changes in anxiety scores over time. The total possible score for the PROMIS for the PROMIS for the PROMIS Anxiety tool ranges from 7 to 35, with higher scores indicating worse outcomes.
Fatigue Inventory Score | At 12 weeks
  Percentage of patients with a 10 percent or greater reduction in brief fatigue inventory score. Fatigue is scored on an 10 points scale (0 to 10), with higher scores indicating worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta K Pal, Principal Investigator — City of Hope Medical Center